CLINICAL TRIAL: NCT04578769
Title: Comparison Study of Conventional Peroral Endoscopic Myotomy (POEM) and Different Modified Procedures of POEM for Achalasia
Brief Title: Assessment of Different Modified POEM for Achalasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Tao Guo, Associated professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUMCH-POEM-1
Record Dates: First submitted 2020-09-26; First posted 2020-10-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Achalasia
Keywords: peroral endoscopic myotomy; Achalasia; thickness of myotomy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional myotomy (Active Comparator): conventional myotomy for achalasia type I or II
  Interventions: Procedure: conventional myotomy
- full-thickness myotomy (Experimental): modified myotomy (full-thickness myotomy) for achalasia type I or II
  Interventions: Procedure: full-thickness myotomy

INTERVENTIONS:
Procedure: conventional myotomy — 1. Initial mucosal incision. After submucosal injection, a reverse T entry incision is made at approximately 10 cm proximal to the gastroesophageal junction (GEJ).
  2. Submucosal tunnel establishment. A submucosal tunnel is created to 2-3 cm distal to the GEJ.
  3. Endoscopic myotomy. A selective circular muscle myotomy is carried out in a proximal to distal direction, from 2 cm distal to the mucosal entry down to 2 cm distal to the GEJ.
  4. Zippered closure of mucosal entry. The mucosal incision is closed using hemostatic clips.
  Other Names: circular myotomy; non-tailored myotomy
  Arms: conventional myotomy
Procedure: full-thickness myotomy — 1. Initial mucosal incision. After submucosal injection, a reverse T entry incision is made at approximately 10 cm proximal to the gastroesophageal junction (GEJ).
  2. Submucosal tunnel establishment. A submucosal tunnel is created to 2-3 cm distal to the GEJ.
  3. Endoscopic myotomy. A selective circular muscle myotomy is carried out in a proximal to distal direction, from 2 cm distal to the mucosal entry down to 4 cm proximal to the GEJ, and a full-thickness muscle myotomy is continually carried out from 4cm proximal to the GEJ down to 2 cm distal to the GEJ.
  4. Zippered closure of mucosal entry. The mucosal incision is closed using hemostatic clips.
  Other Names: modified myotomy
  Arms: full-thickness myotomy

SUMMARY:
The aims of this study is to compare the efficacy and safety of conventional myotomy (circular myotomy) and modified myotomy (full-thickness myotomy) in the treatment of achalasia patients.

DETAILED DESCRIPTION:
Peroral endoscopic myotomy (POEM) is a novel clinical technique used to treat achalasia. The conventional POEM myotomy length averages 8 to 10 cm (4-6 cm in the esophagus, 2-4cm in the LES, 2cm in the cardia & 6-8 cm above and 2 cm below the gastroesophageal junction [GEJ]) for typical achalasia (Chicago classification I, II), with only the inner circular muscle layer incised.

There is still no conclusion on the thickness of muscle bundle dissection recommended during POEM. Selective circular muscle myotomy is designed to avoid gastroesophageal reflux (GER) postoperatively and decrease morbidity during POEM. But one meta-analysis showed that Heller's surgery could keep patients in long-time remission, mainly because of its full-thickness muscle bundle dissection to make sure of persist relaxation of LES. A retrospective study comparing the outcomes of full-thickness and circular muscle myotomy showed no differences in efficacy, GER or adverse events, although the procedural time was shorter in the full thickness myotomy group.

Further randomized controlled trials are warranted to assess the efficacy and safety of different modified myotomy approaches in POEM for patients with achalasia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as achalasia type I or II according to the Chicago Classification Version 4.0, with an Eckardt score >3
* Their age is ≥14years and ≤70 years
* Able to give written consent

Exclusion Criteria:

* undergone previous surgical treatments
* had contra-indication to general anesthesia
* previous surgery of the mediastinum, stomach, or esophagus;
* Pregnant or lactating female
* type III achalasia
* current alcohol or drug addiction, mental retardation, severe congenital or acquired coagulopathy (international normalized ratio >1.6)
* hepatic cirrhosis with or without portal hypertension, eosinophilic esophagitis (biopsies were performed at index endoscopy), or confirmed Barrett's esophagus
* esophageal diverticula or hiatal hernia based on findings from the index barium esophagram, or other conditions that the investigator believed not appropriate for POEM procedure

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Therapeutic success of short term | 6 months after the procedure
  Clinical severity was assessed using the Eckardt score. This score is the sum of the symptom scores for dysphagia, regurgitation, and chest pain (with 0 indicating the absence of symptoms, 1 indicating occasional symptoms, 2 indicating daily symptoms, and 3 indicating symptoms at each meal) and weight loss (with 0 indicating no weight loss, 1 indicating a loss of <5 kg, 2 indicating a loss of 5 to 10 kg, and 3 indicating a loss of >10 kg). The total score ranges from 0 to 12, with higher scores indicating more severe disease symptomatology. (Eckardt, V. Gastroenterology, 1992. 103(6): 1732-8.

SECONDARY OUTCOMES:
Procedure time | During the endoscopic procedure
  The duration of the endoscopic procedures for each patients will be calculated, in minutes, since the mucosal incision until the endoscopic closure of the mucosal entry with the last endoscopic clip.
Pressure changes by high-resolution manometry (HRM) | 6 month after the procedure
  Basal lower esophageal sphincter (LES) pressure, Distal contractile integral (DCI) and integrated relaxation pressure (IRP)
barium esophagogram | 6 month after the procedure
  Barium swallow studies will be done to evaluate the oesophageal emptying at 5 minutes and esophageal distortion
Rate of intra-procedure complications | During the endoscopic procedure
  Complications encountered during the procedure will be noted. (perforation, delayed bleeding, pneumothorax, subcutaneous emphysema, anastomotic leak etc.)
the rate and severity of oesophagitis | 6 months after the procedure
  oesphagitis was identified under esophagogastroduodenoscopy, and was classified according to the Los Angeles Classification
(4) Esophagogastroduodenoscopy (EGD) with the novel Endoscopic Scoring for Achalasia (CARS) | 6-month after the procedure
  Endoscopic evaluation was performed using the Contents, Anatomy, Resistance, and Stasis (CARS) score. This scoring system was developed and validated through video-based reliability assessments and initially demonstrated strong clinical utility for predicting achalasia. The score assigns 0 to 2 points each for Contents, Anatomy, and Resistance at the lower esophageal sphincter, and 1 point for each component of Stasis. The total score ranges from 0 to 8, with higher scores indicating a worse endoscopic outcome.
POEM difficulty evaluation | During the endoscopic procedure
  ① Peroral Endoscopic Myotomy (POEM) difficulty score (PDS). The score consists of five variables: Fibrosis, Oozing, Orientation, Distension of tunnel, and Spastic contractions ("FOODS"). Each variable was arbitrarily weighted equally and assigned values ranging from 0 to 2. The PDS was completed immediately post-procedure in the operating room. The total score ranges from 0 to 10, with higher scores indicating greater technical difficulty. ② bleeding episodes, classified into (1) none to minimal (2) moderate to diffuse
perioperative hospitalization | perioperative period
  perioperative hospitalization length
post-POEM persistent pain | postoperative period
  Post-POEM persistent pain was defined as pain requiring level 2 or 3 analgesics.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Guo, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Gastroenterology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahrilas PJ, Bredenoord AJ, Fox M, Gyawali CP, Roman S, Smout AJ, Pandolfino JE; International High Resolution Manometry Working Group. The Chicago Classification of esophageal motility disorders, v3.0. Neurogastroenterol Motil. 2015 Feb;27(2):160-74. doi: 10.1111/nmo.12477. Epub 2014 Dec 3. PMID 25469569
- [Background] Inoue H, Shiwaku H, Kobayashi Y, Chiu PWY, Hawes RH, Neuhaus H, Costamagna G, Stavropoulos SN, Fukami N, Seewald S, Onimaru M, Minami H, Tanaka S, Shimamura Y, Santi EG, Grimes K, Tajiri H. Statement for gastroesophageal reflux disease after peroral endoscopic myotomy from an international multicenter experience. Esophagus. 2020 Jan;17(1):3-10. doi: 10.1007/s10388-019-00689-6. Epub 2019 Sep 26. PMID 31559513
- [Background] Inoue H, Shiwaku H, Iwakiri K, Onimaru M, Kobayashi Y, Minami H, Sato H, Kitano S, Iwakiri R, Omura N, Murakami K, Fukami N, Fujimoto K, Tajiri H. Clinical practice guidelines for peroral endoscopic myotomy. Dig Endosc. 2018 Sep;30(5):563-579. doi: 10.1111/den.13239. PMID 30022514
- [Background] Wang J, Tan N, Xiao Y, Chen J, Chen B, Ma Z, Zhang D, Chen M, Cui Y. Safety and efficacy of the modified peroral endoscopic myotomy with shorter myotomy for achalasia patients: a prospective study. Dis Esophagus. 2015 Nov-Dec;28(8):720-7. doi: 10.1111/dote.12280. Epub 2014 Sep 12. PMID 25214469
- [Background] Li L, Chai N, Linghu E, Li Z, Du C, Zhang W, Zou J, Xiong Y, Zhang X, Tang P. Safety and efficacy of using a short tunnel versus a standard tunnel for peroral endoscopic myotomy for Ling type IIc and III achalasia: a retrospective study. Surg Endosc. 2019 May;33(5):1394-1402. doi: 10.1007/s00464-018-6414-7. Epub 2018 Sep 5. PMID 30187204
- [Background] Kane ED, Budhraja V, Desilets DJ, Romanelli JR. Myotomy length informed by high-resolution esophageal manometry (HREM) results in improved per-oral endoscopic myotomy (POEM) outcomes for type III achalasia. Surg Endosc. 2019 Mar;33(3):886-894. doi: 10.1007/s00464-018-6356-0. Epub 2018 Jul 27. PMID 30054739
- [Background] Wang XH, Tan YY, Zhu HY, Li CJ, Liu DL. Full-thickness myotomy is associated with higher rate of postoperative gastroesophageal reflux disease. World J Gastroenterol. 2016 Nov 14;22(42):9419-9426. doi: 10.3748/wjg.v22.i42.9419. PMID 27895430
- [Background] Li QL, Chen WF, Zhou PH, Yao LQ, Xu MD, Hu JW, Cai MY, Zhang YQ, Qin WZ, Ren Z. Peroral endoscopic myotomy for the treatment of achalasia: a clinical comparative study of endoscopic full-thickness and circular muscle myotomy. J Am Coll Surg. 2013 Sep;217(3):442-51. doi: 10.1016/j.jamcollsurg.2013.04.033. Epub 2013 Jul 25. PMID 23891074